CLINICAL TRIAL: NCT06974292
Title: The Mass Balance and Biotransformation Study of [14C]VC005 in Chinese Healthy Adult Male Volunteers
Brief Title: The Mass Balance and Biotransformation Study of [14C] VC005 in Chinese Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VC005-105
Record Dates: First submitted 2025-05-06; First posted 2025-05-15 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]VC005 (Experimental)
  Interventions: Drug: [14C]VC005

INTERVENTIONS:
Drug: [14C]VC005 — Take a suspension of 50 mg VC005 ,containing about 120 μCi [14C]VC005, in fasting within 5 minutes

SUMMARY:
This study was designed to evaluate the mass balance and biotransformation after single-dose of [14C]VC005 orally in Chinese healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male adult.
* Age is between 18 and 45, inclusive.
* Weight ≥ 50 kg and Body mass index is between 19 and 26, inclusive.
* Voluntarily to provide informed consent form.
* Willing and able to communicate with investigators and complete the trial according to clinical trial protocol.

Exclusion Criteria:

* Any abnormal and clinical significant findings to physical examination, vital signs, laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, stool routine+occult blood, thyroid function), 12 lead electrocardiogram, chest X-ray (upright position), abdominal ultrasound (liver, gallbladder, pancreas, spleen and kidney), anal directorial rectum examination, and so on.
* Tested positive for any one of the following: HBsAg/HBeAg, Anti-HCV IgG, HIV-Ag/Ab or treponema pallidum antibody (Syphilis) .
* Volunteers who have to work in radioactive conditions in long time, participated in radio-labeled drug clinical trial or had significant radioactive exposure within one year before the trial, more than 2 times of chest/abdominal CT, or more than 3 times of different types of X-ray exam.
* Volunteers are not suitable for this clinical trial, in the opinions of investigators.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion rate of radioactivity in urine | from 0 hour to 216 hours after administration
Cumulative excretion rate of radioactivity in feces | from 0 hour to 216 hours after administration
Total radioactivity | from 0 hour to 216 hours after administration

SECONDARY OUTCOMES:
Adverse events | From signing the ICF until 10 days after the dosing

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Principal Investigator — First Affiliated Hospital of Suzhou Medical College
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China